CLINICAL TRIAL: NCT03666429
Title: Effectiveness of the NoseFrida Compared With Bulb Suction at Relieving Objective Signs of Nasal Obstruction and Reducing Return Visits in Pediatric Patients Presenting to the Emergency Department
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Fridababy (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 181365
Record Dates: First submitted 2018-09-09; First posted 2018-09-11 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Upper Respiratory Tract Infections; Nasal Suction; Return Emergency Department Visits
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Bulb suction (Active Comparator): Patients in this arm will be given bulb suction to treat nasal congestion. This group will contain participants who have used bulb suction in the past.
  Interventions: Device: Bulb suction
- NoseFrida (Experimental): Patients in this arm will be given the NoseFrida to treat nasal congestion. This group will contain participants who will trial the NoseFrida in the emergency department.
  Interventions: Device: NoseFrida

INTERVENTIONS:
Device: Bulb suction — Parents will use the bulb suction on their child in the emergency room then complete a 7 point likert survey.
  Arms: Bulb suction
Device: NoseFrida — Parents will use the NoseFrida in the emergency department and complete a 7 point likert survey.
  Arms: NoseFrida

SUMMARY:
The mainstay of treatment in viral upper and lower respiratory tract disease is airway clearance. Viral respiratory tract infections account for a substantial amount of emergency department (ED) visits, financial and stress burden on caregivers. In addition, they also account for a large number of ED return visits. While airway clearance is considered a mainstay of treatment the pragmatic effectiveness of various devices remain unstudied in patients who are discharged from the ED.

The objectives of this study are to compare the pragmatic effectiveness of two commonly used suction devices the NoseFrida and bulb suction and to provide a descriptive analysis on 72 hour return to ED rates and readmission rates. Patients will be enrolled October 15, 2018 to October 15, 2019 or until NoseFrida supplies are depleted. Fridababy will supply 500 NoseFrida devices and replacement filters. Patients aged 1 day to 24 months presenting Vanderbilt Childrens ED with symptoms of nasal congestion or bronchiolitis who require suctioning and will be discharged from the ED will be approached for enrollment. Exclusion criteria include no upper airway abnormalities or previously enrolled in study. The study design is a prospective and retrospective observational study. We anticipate about 500 patients to be enrolled in this study. Families will then be approached for consent to participate. Caregiver will fill out a data collection form then be instructed on how to use the NoseFrida. Next, family with trial it on their child while in the ED. Caregivers will then fill out a 7 point Likert survey on both the bulb suction and NoseFrida device. The family will go home with this device and a set of replacement filters and instructed to suction their child as needed. The primary investigator (PI) will then complete a 72 hour chart review to determine the number of return to ED visits and readmission rates. To compare ED returns with retrospective data, KSP will conduct a review of the business objects database using ICD9 codes specific for viral respiratory tract infections over the past 3 years to determine a control return ED visit rate. Data will be compared using a paired T-test. If data is not normally distributed we will use a Wilcoxon signed-rank test. We will also use a multivariable logistic model to examine associations adjusted for age and illness severity.

DETAILED DESCRIPTION:
Background The mainstay of treatment in viral upper and lower respiratory tract disease is airway clearance. Viral respiratory tract infections account for a substantial amount of emergency department (ED) visits, financial and stress burden on caregivers. In addition, they also account for a large number of ED return visits. While airway clearance is considered a mainstay of treatment the pragmatic effectiveness of various devices remain unstudied in patients who are discharged from the ED.

Hypothesis:

There is no difference between the NoseFrida and the bulb suction at relieving objective signs of nasal obstruction or return ED visits.

Study Objective:

1. To compare the use of the NoseFrida device with a retrospective control (bulb suction) to determine if there is a decrease in the number of ED return visits.
2. To provide evidence based recommendations on the pragmatic effectiveness of two commonly used suction devices.
3. To provide a descriptive analysis on 72 hour return to ED rates and readmission rates.

Methods:

The study design is a prospective and retrospective observational study. We anticipate about 500 patients to be enrolled in this study. Patients who present to Vanderbilt Childrens Emergency Department will be identified by key study personnel (KSP) based on inclusion and exclusion criteria. Families will then be approached for consent to participate. Caregiver will fill out a data collection form then be instructed on how to use the NoseFrida. Next, family with trial it on their child while in the ED. Caregivers will then fill out a 7 point Likert survey on both the bulb suction and NoseFrida device. The family will go home with this device and a set of replacement filters and instructed to suction their child as needed. The primary investigator (PI) will then complete a 72 hour chart review to determine the number of return to ED visits and readmission rates. The family will keep the suction device at the completion of the study. To compare ED returns with retrospective data, KSP will conduct a review of the business objects database using ICD9 codes specific for viral respiratory tract infections over the past 3 years to determine a control return ED visit rate. Data will be compared using a paired T-test. If data is not normally distributed we will use a Wilcoxon signed-rank test. We will also use a multivariable logistic model to examine associations adjusted for age and illness severity. Fridababy will provide supplies needed for the study, however the company will not have access to the raw data or PHI. Once the results are published in a scientific journal, then Fridababy will have access to the results.

ELIGIBILITY:
Inclusion Criteria:

1. Age 1 day-24 months presenting to the ED with a complaint of nasal congestion or symptoms of bronchiolitis who require suctioning.
2. Parent/guardian has used a bulb suction device in the past.
3. This is the first presentation to Vanderbilt Childrens Emergency Department for current illness.
4. Patient will be discharged from the emergency room.
5. Parent/Guardian is able to read English.

Exclusion Criteria:

1. No upper airway abnormalities, i.e. cleft palate or choanal atresia.
2. Previously enrolled in study.

Ages: 1 Day to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Parental satisfaction | at baseline
  Measured on a 7 point Likert scale from 1 to 7 with 7 being strongly agree

CONTACTS AND LOCATIONS:
Overall Officials: Donald Arnold, M.D., Study Chair — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Childrens Emergency Department, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No